CLINICAL TRIAL: NCT01474993
Title: Sulforaphane-rich Broccoli Sprout Extract for Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Andrew Zimmerman (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor-Investigator, Andrew Zimmerman, Pediatric Neurologist, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011P002221
Record Dates: First submitted 2011-11-08; First posted 2011-11-18 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): inactive placebo.
  Interventions: Drug: Placebo
- Interventional (Experimental): sulforaphane-rich Broccoli Sprout Extract.
  Interventions: Drug: Sulforaphane-rich Broccoli Sprout Extract

INTERVENTIONS:
Drug: Sulforaphane-rich Broccoli Sprout Extract — 30 subjects will be randomly selected to receive sulforaphane-rich Broccoli Sprout Extract. The medication will be supplied and dispensed as No.1 size gelcaps (each gelcap containing ~ 250 mg sulforaphane rich Broccoli Sprout Extract, equivalent to ~ 50 µmol of sulforaphane). The dosage of sulforaphane will depend on subject's body weight:
  1. Subjects with body weight less than 101 lbs will receive ~ 50 micromol sulforaphane per day (1 gelcap to be taken once a day)
  2. Subjects with body weight 101 lbs to 199 lbs will receive ~ 100 micromol sulforaphane per day (2 gelcaps to be taken once a day)
  3. Subjects with bidy weight > 199 lbs will receive ~ 150 micromol sulforaphane per day (3 gelcaps to be taken once a day)
  Arms: Interventional
Drug: Placebo — 15 subjects will be randomly selected to receive inactive placebo (Gelcaps identical in appearance to that of active medication and containing microcrystalline cellulose)
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to answer whether there is evidence of measurable effects on social responsiveness (primary outcome) and other behavioral symptoms after treatment of autistic male adolescents and adults with orally administered sulforaphane-rich Broccoli Sprout Extract (efficacy). The secondary objectives of this study are to answer whether treatment of male adolescents and adults with autism using orally administered sulforaphane-rich Broccoli Sprout Extract within a specified dose range is safe (toxicity); treatment with sulforaphane-rich Broccoli Sprout Extract is well tolerated (side effects and adverse events); key cellular biomarkers support the hypothesized mechanisms (proof of principle).

DETAILED DESCRIPTION:
Behavioral improvements occur transiently during febrile illnesses in autism, and include decreased repetitive behaviors and improved speech. These changes have been recorded in 38% of autistic children in a clinical survey and 83% in an observational study, respectively. The cellular basis for this "fever effect" is unknown but is likely to involve heat shock proteins (HSP) and cellular stress responses (CSR) that lead to changes in synaptic function and network connectivity.

Sulforaphane (1-isothiocyanato-4R- (methylsulfinyl)butane) is an isothiocyanate that is delivered by lyophilized extracts of 3-day-old broccoli sprouts. Broccoli sprouts are widely consumed as a food item all over the world by very large numbers of individuals, without any reports of adverse effects. Our preliminary work in vitro shows that sulforaphane stimulates HSP and mitochondrial biogenesis in several genetic disorders.

This study of sulforaphane-rich Broccoli Sprout Extract in autism is a randomized, double-blinded, placebo-controlled, phase II single site trial, designed to ensure safety and obtain efficacy data, with a focus on changes in social responsiveness, a core feature of autism. Its hybrid design, incorporating double masking, placebo control, and randomization, enhances the robustness of early outcome data. The study duration will be 2 years. Recruitment of subjects will be 50% by 8 months and complete by 14 months. All subjects in the study will be followed for 22 weeks. Treatment (18 weeks) will be started as patients are entered into the study and receive baseline testing. All treatment will be completed by 20 months and data analysis and presentation of results by 24 months.

Forty-five male adolescents (13-18 years) and adults (19-30 years) with autism will be randomly assigned to receive either sulforaphane-rich Broccoli Sprout Extract (n = 30) or placebo (n = 15). The 2:1 randomization schedule will be produced by the study statistician using permuted random blocks and stratification by history of positive behavioral effects of fever. Treatment assignments will be performed by the research pharmacy at MGH. Females will be excluded for homogeneity of the sample and because males have higher incidence of autism than females (4:1). We will seek to enroll up to 50% of the subjects having a history of positive behavioral effects of fever, which will be recorded from caregivers' recall of incidents and graded on the CGI-Improvement (CGI-I) 7-point scale.

There will be in total 7 study visits for each subject: the screening visit, enrollment visit, a blood draw visit at 24 hours after the first dose of study medication (for mitochondrial/heat shock protein analysis), 4 week (follow-up) visit, 10 week (follow-up) visit, 18 week visit (last treatment visit), and the final closeout visit one month after the study drug stops (22 weeks). Even though the treatment will stop at 18 weeks, we will follow subjects for additional 4 weeks after study medication stops (the 22 week visit) to ensure safety after study drug stops. Additional visits may be conducted in case any side effects are reported at any stage of the study.

ELIGIBILITY:
Inclusion Criteria:

* Autism diagnosis. Quantitative autism traits and severity for diagnosis of autism will be assessed using the ADOS-G (Modules 1-4 and Severity), Social Responsiveness Scale (SRS; child and adult forms), Clinical Global Impression-Severity (CGI-S) and Aberrant Behavior Checklist-Withdrawal subscale (ABC-W).

Exclusion Criteria:

* Absence of a parent or legal guardian and consent
* Unavailability for all visits and adherence to study regimen
* Seizure within 2 years of screening
* Impaired renal function (serum creatinine > 1.2 mg/dl), impaired hepatic function (AST/ALT > 2x upper limit of normal), impaired thyroid function (TSH outside normal limits)
* Current infection or treatment with antibiotics; AND
* Chronic medical disorder (e.g., cardiovascular disease, stroke or diabetes) or major surgery within 3 months prior to enrollment.
* A diagnosis of autism spectrum disorder other than autism, for example, Asperger's, PDD-NOS etc.

Ages: 13 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W. Zimmerman, M.D., Principal Investigator — UMass Medical School
Locations (1):
- Lurie Center for Autism, MassGeneral Hospital for Children, Lexington, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-four study participants were initially enrolled in the study from January 2011 to July 2013 at Lurie Center for Autism.
Groups:
- Placebo: 15 participants were randomized to placebo (Gelcaps identical in appearance to that of active medication and containing microcrystalline cellulose).One participant in placebo group dropped out before starting study drug. 14 participants completed the study.
- Sulforaphane-rich Broccoli Sprout Extract: 29 subjects were randomized to receive sulforaphane-rich Broccoli Sprout Extract. Of these, 2 were lost to follow up and 1 discontinued intervention. 26 sulforaphane participants completed the study.
  Sulforaphane-rich Broccoli Sprout Extract: The medication was supplied and dispensed as No.1 size gelcaps (each gelcap containing ~ 250 mg sulforaphane rich Broccoli Sprout Extract, equivalent to ~ 50 µmol of sulforaphane). The dosage of sulforaphane depended on subject's body weight:
  1. Subjects with body weight less than 101 lbs will receive ~ 50 micromol sulforaphane per day (1 gelcap to be taken once a day)
  2. Subjects with body weight 101 lbs to 199 lbs will receive ~ 100 micromol sulforaphane per day (2 gelcaps to be taken once a day)
  3. Subjects with bidy weight > 199 lbs will receive ~ 150 micromol sulforaphane per day (3 gelcaps to be taken once a day)
Period: Overall Study
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Started | 15 | 29
Completed | 14 | 26
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 15 participants were randomized to placebo.
- Sulforaphane-rich Broccoli Sprout Extract: 29 subjects were randomized to receive sulforaphane.
- Total: Total of all reporting groups
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract | Total
Number analyzed (Participants) | 15 | 29 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.6 (3.5) | 17.9 (3.9) | 17.4 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 15 | 29 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 13 | 26 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 29 | 44
Aberrant Behavior Checklist total score [Mean (Standard Deviation); unit: units on a scale] — The Aberrant Behavior Checklist has 58 questions rated by parents or teachers on a scale of 0 to 3, where a score of "0" for particular behavior is not a problem at all, "1" indicates that the behavior is a problem but slight in degree, "2" indicates that the problem is moderately serious, and "3" indicates that the problem is severe in degree. The possible ABC scores may range from 0 to 174, where higher values represent the worse outcome.
  units on a scale | 60 (23.2) | 63.6 (25.3) | 62.3 (24.4)
Social Responsiveness Scale total score [Mean (Standard Deviation); unit: units on a scale] — The Social Responsiveness Scale is a parent- and/or teacher-reported 65 question scale. Each question on the scale inquires about an observed aspect of reciprocal social behavior that is rated on the scoring sheet on a scale from "0" to "3", where 0 is best possible behavior and 3 is the worst possible behavior. The total SRS score may range from 0 to 195 where higher values represent the worse outcome.
  units on a scale | 120.1 (16.6) | 122.2 (24.1) | 121.5 (21.6)
OACIS-S general level of autism score [Mean (Standard Deviation); unit: units on a scale] — This question on the Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) inquires about the overall level of autism. The question is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
  units on a scale | 4.53 (0.74) | 4.38 (0.56) | 4.43 (0.62)
OACIS-S social interaction score [Mean (Standard Deviation); unit: units on a scale] — This question on the Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) inquires about social interaction impairment. The question is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
  units on a scale | 4.80 (1.01) | 4.51 (0.69) | 4.61 (0.81)
OACIS-S aberrant behavior score [Mean (Standard Deviation); unit: units on a scale] — This question on the Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) inquires aberrant behaviors (such as aggressions etc.). The question is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
  units on a scale | 4.20 (1.37) | 4.21 (0.86) | 4.20 (1.05)
OACIS-S repetitive behavior score [Mean (Standard Deviation); unit: units on a scale] — This question on the Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) inquires about repetitive/ritualistic behaviors. The question is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
  units on a scale | 4.13 (0.83) | 4.14 (0.74) | 4.13 (0.77)
OACIS-S verbal communication score [Mean (Standard Deviation); unit: units on a scale] — This question on the Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) inquires about impairment of verbal communication skills. The question is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
  units on a scale | 4.53 (1.36) | 4.45 (0.95) | 4.48 (1.09)
OACIS-S nonverbal communication score [Mean (Standard Deviation); unit: units on a scale] — This question on the Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) inquires about impairment of non-verbal communication skills. The question is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
  units on a scale | 4.27 (0.96) | 4.10 (0.72) | 4.16 (0.81)
OACIS-S hyperactivity/inattention score [Mean (Standard Deviation); unit: units on a scale] — This question on the Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) inquires about severity of hyperactivity and inattentiveness. The question is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
  units on a scale | 4.40 (0.91) | 4.10 (0.90) | 4.20 (0.90)
OACIS-S anxiety score [Mean (Standard Deviation); unit: units on a scale] — This question on the Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) inquires about severity of anxiety. The question is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
  units on a scale | 4.33 (1.23) | 4.17 (0.71) | 4.23 (0.91)
OACIS-S sensory sensitivity score [Mean (Standard Deviation); unit: units on a scale] — This question on the Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) inquires about severity of sensory sensitivities. The question is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
  units on a scale | 4.40 (0.74) | 4.07 (0.65) | 4.18 (0.69)
OACIS-S restricted interests score [Mean (Standard Deviation); unit: units on a scale] — This question on Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) inquires about restricted and narrow interests of the patient. The question is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
  units on a scale | 4.33 (0.72) | 4.41 (0.63) | 4.38 (0.65)
Hematology: Red Blood Cell (RBC) counts [Mean (Standard Deviation); unit: *10^6 cells/µL] | 5.1 (0.3) | 5.2 (0.5) | 5.2 (0.4)
Hematology: White Blood Cell (WBC) counts [Mean (Standard Deviation); unit: *10^03 cells/µL] | 6.9 (2.3) | 6.8 (1.7) | 6.8 (1.9)
Hematology: platelet counts [Mean (Standard Deviation); unit: *10^03 cells/µL] | 245.5 (47.8) | 251.5 (55.5) | 249.6 (52.6)
Blood chemistry: serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.8 (0.1) | 0.8 (0.1) | 0.8 (0.1)
Blood Chemistry: Serum glutamic oxaloacetic transaminase (SGOT) [Mean (Standard Deviation); unit: U/L] | 22.8 (6.4) | 22.6 (8.6) | 22.7 (7.9)
Blood Chemistry: Serum glutamic pyruvic transaminase (SGPT) [Mean (Standard Deviation); unit: U/L] | 18.3 (6.1) | 30.0 (20.6) | 26.3 (18.1)
Blood chemistry: Thyroid Stimulating Hormone (TSH) [Mean (Standard Deviation); unit: uIU/mL] | 1.6 (0.9) | 2.0 (2.1) | 1.9 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Screening/Baseline in Social Responsiveness Scale (SRS) at 4 Weeks, 10 Weeks, 18 Weeks and 22 Weeks
Description: The Social Responsiveness Scale is a parent- and/or teacher-reported 65 question scale. Each question on the scale inquires about an observed aspect of reciprocal social behavior that is rated on the scoring sheet on a scale from "0" to "3", where 0 is best possible behavior and 3 is the worst possible behavior. The total SRS score may range from 0 to 195 where higher values represent the worse outcome.
  For the purposes of this study, SRS scores were obtained at both screening (the day study participants were first seen and consent obtained) and the baseline visits (the day study medication was first started, within a month of the screening visit). The screening and baseline scores were then averaged and these average SRS scores were used to calculate the change in scores at 4 weeks, 10 weeks, 18 weeks and 22 weeks respectively.
Time Frame: 4 weeks, 10 weeks, 18 weeks and 22 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Patients were treated for 18 weeks (from the second [baseline] visit until the 18 week visit). The placebo was supplied and dispensed as no.1 size gel caps (each gel cap containing microcrystalline cellulose) identical in size, appearance and color to capsules containing sulforaphane. The dosage of placebo was based on the patient's body weight: 1 gel cap per day for patients with weight ≤ 100 lbs; 2 gel caps per day for patients with weight 101 - 199 lbs; 3 gel caps per day for patients with weight ≥ 200 lbs. Route of administration: oral. Frequency of administration: once a day.
- Sulforaphane-rich Broccoli Sprout Extract: Patients were treated for 18 weeks (from the second [randomization] visit until the 18 week visit). Sulforaphane was supplied and dispensed as no.1 size gel caps (each gel cap containing ~ 250 mg Sulforaphane rich Broccoli Sprout Extract, equivalent to ~ 50 µmol of Sulforaphane). The dosage of Sulforaphane was based on the patient's body weight: ~50 µmol Sulforaphane (1 gel cap per day) for patients with weight ≤ 100 lbs; ~100 µmol Sulforaphane (2 gel caps per day) for patients with weight 101 - 199 lbs; ~150 µmol Sulforaphane (3 gel caps per day) for patients with weight ≥ 200 lbs. Route of administration: oral. Frequency of administration: once a day.
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Number analyzed (Participants) | 14 | 26
units on a scale
  Change from screening/baseline at 4 weeks | -7.79 (3.09) | -14.76 (3.79)
  Change from screening/baseline at 10 weeks | -1.38 (3.72) | -14.48 (5.72)
  Change from screening/baseline at 18 weeks | -2.0 (3.46) | -20.40 (4.54)
  Change from screening/baseline at 22 weeks | -6.67 (3.82) | -7.03 (4.20)

2. Secondary Outcome: Change From Screening/Baseline in Aberrant Behavior Checklist (ABC) at 4 Weeks, 10 Weeks, 18 Weeks and 22 Weeks
Description: The Aberrant Behavior Checklist has 58 questions rated by parents or teachers on a scale of 0 to 3, where a score of "0" for particular behavior is not a problem at all, "1" indicates that the behavior is a problem but slight in degree, "2" indicates that the problem is moderately serious, and "3" indicates that the problem is severe in degree. The possible ABC scores may range from 0 to 174, where higher values represent the worse outcome.
  For the purposes of this study, ABC scores were obtained at both screening (the day study participants were first seen and consent obtained) and the baseline visits (the day study medication was first started, within a month of the screening visit). The screening and baseline scores were then averaged and these average ABC scores were used to calculate the change in scores at 4 weeks, 10 weeks, 18 weeks and 22 weeks respectively.
Time Frame: 4 weeks, 10 weeks, 18 weeks, 22 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Number analyzed (Participants) | 14 | 26
units on a scale
  Change from screening/baseline at 4 weeks | 0.77 (1.84) | -12.69 (4.17)
  Change from screening/baseline at 10 weeks | 3.31 (3.50) | -19.61 (5.95)
  Change from screening/baseline at 18 weeks | -2.0 (4.59) | -21.44 (4.34)
  Change from screening/baseline at 22 weeks | -1.83 (6.60) | -10.72 (5.07)

3. Secondary Outcome: Ohio Autism Clinical Global Impression Scale - Severity (OACIS-S) Scale at 4 Weeks, 10 Weeks, 18 Weeks and 22 Weeks
Description: OACIS-S is a 10 domain scale that requires the clinician to rate the severity of the patient's autism symptoms at the time of assessment. The 10 domains cover different aspects of patients' behavior, including global autism severity, social interaction, aberrant behavior, repetitive or ritualistic behaviors, verbal communication, non-verbal communication, hyperactivity/inattention, anxiety, sensory sensitivities and restricted/narrow interests.
  Each domain is rated on a scale of 1 to 7 where 1 is normal, 2 is some symptoms sometimes affecting individual and family, 3 is mild symptoms affecting individual daily and sometimes family, 4 is moderate symptoms affecting individual and family daily, 5 is marked symptoms affecting individual daily and sometimes family, 6 is severe symptoms affecting individual daily and sometimes family, and 7 is severe symptoms affecting individual and family daily.
Time Frame: 4 weeks, 10 weeks, 18 weeks, 22 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Number analyzed (Participants) | 14 | 26
units on a scale
  OACIS-S general level of autism 4 weeks | 4.36 (0.84) | 4.38 (0.80)
  OACIS-S general level of autism 10 weeks | 4.43 (0.85) | 4.31 (0.74)
  OACIS-S general level of autism 18 weeks | 4.50 (0.76) | 4.42 (0.70)
  OACIS-S general level of autism 22 weeks | 4.70 (0.82) | 4.50 (0.89)
  OACIS-S social interaction 4 weeks | 4.50 (1.16) | 3.77 (0.99)
  OACIS-S social interaction 10 weeks | 4.57 (1.28) | 3.46 (1.03)
  OACIS-S social interaction 18 weeks | 4.71 (1.27) | 3.46 (1.14)
  OACIS-S social interaction 22 weeks | 5.0 (1.41) | 4.60 (1.05)
  OACIS-S aberrant behavior 4 weeks | 4.36 (1.34) | 3.73 (1.25)
  OACIS-S aberrant behavior 10 weeks | 4.29 (1.07) | 3.27 (1.12)
  OACIS-S aberrant behavior 18 weeks | 4.43 (1.22) | 3.19 (1.23)
  OACIS-S aberrant behavior 22 weeks | 4.90 (1.60) | 4.35 (1.63)
  OACIS-S repetitive behavior 4 weeks | 3.86 (1.10) | 4.08 (0.98)
  OACIS-S repetitive behavior 10 weeks | 4.14 (0.86) | 3.62 (1.33)
  OACIS-S repetitive behavior 18 weeks | 4.14 (0.77) | 3.69 (1.19)
  OACIS-S repetitive behavior 22 weeks | 4.30 (0.82) | 4.55 (0.89)
  OACIS-S verbal communication 4 weeks | 4.43 (1.70) | 3.73 (1.25)
  OACIS-S verbal communication 10 weeks | 4.21 (1.85) | 3.73 (1.08)
  OACIS-S verbal communication 18 weeks | 4.71 (1.33) | 3.54 (1.10)
  OACIS-S verbal communication 22 weeks | 5.20 (1.32) | 4.80 (1.15)
  OACIS-S non-verbal communication 4 weeks | 4.29 (0.99) | 3.85 (1.01)
  OACIS-S non-verbal communication 10 weeks | 4.23 (1.01) | 3.73 (1.04)
  OACIS-S non-verbal communication 18 weeks | 4.43 (0.94) | 3.69 (1.12)
  OACIS-S non-verbal communication 22 weeks | 4.40 (1.08) | 4.25 (1.02)
  OACIS-S hyperactivity 4 weeks | 4.36 (1.01) | 3.50 (1.14)
  OACIS-S hyperactivity 10 weeks | 4.07 (1.27) | 3.54 (0.90)
  OACIS-S hyperactivity 18 weeks | 4.29 (1.07) | 3.58 (1.17)
  OACIS-S hyperactivity 22 weeks | 4.20 (1.32) | 4.25 (1.12)
  OACIS-S anxiety 4 weeks | 4.21 (0.89) | 3.81 (0.98)
  OACIS-S anxiety 10 weeks | 4.43 (0.94) | 3.69 (1.01)
  OACIS-S anxiety 18 weeks | 4.36 (1.01) | 3.85 (1.01)
  OACIS-S anxiety 22 weeks | 4.50 (1.08) | 4.20 (0.89)
  OACIS-S sensory sensitivity 4 weeks | 4.36 (0.50) | 4.08 (0.74)
  OACIS-S sensory sensitivity 10 weeks | 4.43 (0.65) | 4.00 (0.75)
  OACIS-S sensory sensitivity 18 weeks | 4.57 (0.51) | 4.04 (1.00)
  OACIS-S sensory sensitivity 22 weeks | 4.60 (0.52) | 4.20 (1.11)
  OACIS-S restricted interests 4 weeks | 4.07 (0.73) | 4.27 (0.96)
  OACIS-S restricted interests 10 weeks | 4.00 (0.96) | 3.92 (0.98)
  OACIS-S restricted interests 18 weeks | 4.21 (0.89) | 3.92 (1.09)
  OACIS-S restricted interests 22 weeks | 4.50 (0.97) | 4.55 (1.10)

4. Secondary Outcome: Ohio Autism Clinical Impressions Scale - Improvement (OACIS-I) (or CGI-I Scores) Scores at 4 Weeks, 10 Weeks, 18 Weeks and 22 Weeks
Description: The Ohio Autism Clinical Impressions Improvement Scale (OACIS-I) is a 10 domain scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to the baseline state at the beginning of the intervention. The 10 domains cover different aspects of patients' behavior, including global autism severity, social interaction, aberrant behavior, repetitive or ritualistic behaviors, verbal communication, non-verbal communication, hyperactivity/inattention, anxiety, sensory sensitivities and restricted/narrow interests.
  Each domain is rated on a scale of 1 to 7, where "1" is very much improved; "2" is much improved; "3" is minimally improved; "4" is no change; "5" is minimally worse; "6" is much worse; or "7" is very much worse.
Time Frame: 4 weeks, 10 weeks, 18 weeks, 22 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Number analyzed (Participants) | 14 | 26
units on a scale
  OACIS-I general level of autism 4 weeks | 4.14 (0.53) | 4.04 (0.20)
  OACIS-I general level of autism 10 weeks | 3.86 (0.36) | 3.88 (0.33)
  OACIS-I general level of autism 18 weeks | 3.93 (0.27) | 3.81 (0.40)
  OACIS-I general level of autism 22 weeks | 4.0 (0) | 3.92 (0.27)
  OACIS-I social interaction 4 weeks | 3.71 (0.61) | 3.38 (0.85)
  OACIS-I social interaction 10 weeks | 3.79 (0.58) | 3.08 (0.89)
  OACIS-I social interaction 18 weeks | 3.92 (0.47) | 3.08 (1.02)
  OACIS-I social interaction 22 weeks | 4.1 (0.32) | 4.2 (0.77)
  OACIS-I aberrant behavior 4 weeks | 3.86 (0.66) | 3.42 (0.99)
  OACIS-I aberrant behavior 10 weeks | 3.79 (0.58) | 2.96 (1.0)
  OACIS-I aberrant behavior 18 weeks | 3.93 (0.73) | 2.88 (0.99)
  OACIS-I aberrant behavior 22 weeks | 4.2 (0.64) | 4.1 (1.12)
  OACIS-I repetitive behavior 4 weeks | 3.71 (0.61) | 3.81 (0.57)
  OACIS-I repetitive behavior 10 weeks | 4 (0) | 3.35 (0.89)
  OACIS-I repetitive behavior 18 weeks | 4 (0.39) | 3.42 (0.86)
  OACIS-I repetitive behavior 22 weeks | 4.1 (0.32) | 4.25 (0.55)
  OACIS-I verbal communication 4 weeks | 3.57 (0.76) | 3.15 (0.92)
  OACIS-I verbal communication 10 weeks | 3.36 (0.84) | 3.16 (0.83)
  OACIS-I verbal communication 18 weeks | 3.86 (0.53) | 2.96 (0.92)
  OACIS-I verbal communication 22 weeks | 4 (0.47) | 4.15 (0.59)
  OACIS-I non-verbal communication 4 weeks | 3.93 (0.27) | 3.69 (0.62)
  OACIS-I non-verbal communication 10 weeks | 3.92 (0.28) | 3.58 (0.76)
  OACIS-I non-verbal communication 18 weeks | 4.07 (0.27) | 3.54 (0.764)
  OACIS-I non-verbal communication 22 weeks | 4 (0) | 4 (0.46)
  OACIS-I hyperactivity 4 weeks | 4 (0) | 3.42 (0.90)
  OACIS-I hyperactivity 10 weeks | 3.71 (0.61) | 3.46 (0.81)
  OACIS-I hyperactivity 18 weeks | 3.93 (0.62) | 3.5 (0.86)
  OACIS-I hyperactivity 22 weeks | 3.8 (0.42) | 4.05 (0.69)
  OACIS-I anxiety 4 weeks | 4 (0) | 3.65 (0.74)
  OACIS-I anxiety 10 weeks | 4.21 (0.43) | 3.54 (0.81)
  OACIS-I anxiety 18 weeks | 4.14 (0.36) | 3.69 (0.27)
  OACIS-I anxiety 22 weeks | 4.2 (0.42) | 4 (0.46)
  OACIS-I sensory sensitivity 4 weeks | 3.86 (0.36) | 3.85 (0.54)
  OACIS-I sensory sensitivity 10 weeks | 3.93 (0.27) | 3.77 (0.51)
  OACIS-I sensory sensitivity 18 weeks | 4.07 (0.27) | 3.81 (0.63)
  OACIS-I sensory sensitivity 22 weeks | 4 (0) | 4 (0.65)
  OACIS-I restricted interests 4 weeks | 3.86 (0.53) | 3.81 (0.49)
  OACIS-I restricted interests 10 weeks | 3.79 (0.43) | 3.46 (0.71)
  OACIS-I restricted interests 18 weeks | 4 (0) | 3.46 (0.86)
  OACIS-I restricted interests 22 weeks | 4.1 (0.32) | 4.05 (0.83)

5. Secondary Outcome: Liver Function Tests [Serum Glutamic Oxaloacetic Transaminase (SGOT) and Serum Glutamic Pyruvic Transaminase (SGPT)] at 4 Weeks, 18 Weeks and 22 Weeks
Time Frame: 4 weeks, 18 weeks, 22 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Number analyzed (Participants) | 14 | 26
U/L
  SGOT 4 weeks | 27.6 (9.4) | 23.8 (8.3)
  SGOT 18 weeks | 22.5 (9.2) | 22.5 (5.4)
  SGOT 22 weeks | 21.8 (4.1) | 25.4 (13.1)
  SGPT 4 weeks | 25.1 (16.8) | 23.8 (8.3)
  SGPT 18 weeks | 22.2 (20.1) | 31.1 (20.7)
  SGPT 22 weeks | 21 (10.4) | 37.7 (33)

6. Secondary Outcome: Renal Function Tests (Serum Creatinine) at 4 Weeks, 18 Weeks and 22 Weeks
Time Frame: 4 weeks, 18 weeks, 22 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Number analyzed (Participants) | 14 | 26
mg/dL
  Serum Creatinine at 4 weeks | 0.8 (0.1) | 0.8 (0.1)
  Serum Creatinine at 18 weeks | 0.8 (0.1) | 0.8 (0.1)
  Serum Creatinine at 22 weeks | 0.8 (0.1) | 0.8 (0.1)

7. Secondary Outcome: Thyroid Stimulating Hormone (TSH) at 4 Weeks, 18 Weeks and 22 Weeks
Time Frame: 4 weeks, 18 weeks, 22 weeks
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Number analyzed (Participants) | 14 | 26
uIU/mL
  TSH 4 weeks | 1.8 (1.0) | 1.8 (0.8)
  TSH 18 weeks | 1.5 (0.6) | 1.9 (1.1)
  TSH 22 weeks | 1.2 (0.58) | 1.7 (0.7)

8. Secondary Outcome: Red Blood Cell (RBC) Count at 4 Weeks, 18 Weeks and 22 Weeks
Time Frame: 4 weeks, 18 weeks, 22 weeks
Measure: Mean (Standard Deviation); unit: *10^6 cells/µL
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Number analyzed (Participants) | 14 | 26
*10^6 cells/µL
  RBC count at 4 weeks | 5.13 (0.36) | 5.11 (0.36)
  RBC count at 18 weeks | 5.03 (0.38) | 5.13 (0.40)
  RBC count at 22 weeks | 5.12 (0.37) | 5.04 (0.38)

9. Secondary Outcome: White Blood Cell (WBC) Count at 4 Weeks, 18 Weeks and 22 Weeks
Time Frame: 4 weeks, 18 weeks, 22 weeks
Measure: Mean (Standard Deviation); unit: *10^3 cells/µL
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Number analyzed (Participants) | 14 | 26
*10^3 cells/µL
  WBC count at 4 weeks | 6.63 (1.91) | 6.32 (1.56)
  WBC count at 18 weeks | 6.33 (1.71) | 5.94 (1.63)
  WBC count at 22 weeks | 6.12 (1.45) | 6.18 (1.84)

10. Secondary Outcome: Platelet Count at 4 Weeks, 18 Weeks and 22 Weeks
Time Frame: 4 weeks, 18 weeks, 22 weeks
Measure: Mean (Standard Deviation); unit: *10^3 cells/µL
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Number analyzed (Participants) | 14 | 26
*10^3 cells/µL
  Platelet count at 4 weeks | 242.1 (48.1) | 235.0 (38.3)
  Platelet count at 18 weeks | 236.8 (44.8) | 237.1 (45.2)
  Platelet count at 22 weeks | 218.1 (49.2) | 255.0 (52.2)

11. Secondary Outcome: Change From Screening and Baseline in Urinary Isoprostane F2α-VI Levels at 24 Hours After First Dose, at 4 Weeks, 10 Weeks, 18 Weeks and 22 Weeks
Description: *Due to lack of resources, only the results on change from screening at the final intervention visit (18 weeks) are reported.
Time Frame: Screening, baseline, 24 hours after first dose of study medication, 4 weeks, 10 weeks, 18 weeks, 22 weeks
Population: *Due to lack of resources and issues with participant compliance, only the results on change from screening at the final intervention visit (18 weeks) in 13 placebo recipients are reported.
Measure: Mean (Standard Deviation); unit: pG/mL
Arm/Group | Placebo | Interventional
Number analyzed (Participants) | 13 | 26
pG/mL | 0.007 (0.11) | 0.017 (0.09)

12. Secondary Outcome: Change From the Screening Visit in Heat Shock Protein Gene Expression (Relative Maximum Gene Expression) at 24 Hours After First Dose, 18 Weeks and 22 Weeks
Description: Due to lack of resources, only the results on change from screening at the final intervention visit (18 weeks) are reported.
Time Frame: Screening, 24 hours after first dose of study medication, 18 weeks, 22 weeks
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | Placebo | Interventional
Number analyzed (Participants) | 14 | 26
fold change | -0.116 (0.037) | -0.0008 (0.014)

ADVERSE EVENTS:
Time Frame: 22 weeks
Groups:
- Placebo: 15 participants were randomized to placebo. One participant in placebo group dropped out before starting study drug. 14 participants completed the study and were analyzed.
- Sulforaphane-rich Broccoli Sprout Extract: 29 subjects were randomized to receive sulforaphane-rich Broccoli Sprout Extract. Of these, 2 were lost to follow up and 1 discontinued intervention. 26 sulforaphane participants completed the study and were analyzed.
Arm/Group | Placebo | Sulforaphane-rich Broccoli Sprout Extract
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/26
Other Adverse Events (participants affected / at risk) | 4/14 | 5/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Sulforaphane-rich Broccoli Sprout Extract (N=26)
Vomiting (Gastrointestinal disorders) | 1 | 5
Increased aggressions (Psychiatric disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Increased Flatulence (Gastrointestinal disorders) | 2 | 4
Increased irritability (Psychiatric disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 2 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 3
Fever (General disorders) | 1 | 3
Headache (Nervous system disorders) | 1 | 3
Seasonal allergy exacerbation (General disorders) | 0 | 3
Seizures (Nervous system disorders) | 0 (0) | 2 (2)
Increased stubbornness (Psychiatric disorders) | 0 | 2
Insomnia (General disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Increased agitation (Psychiatric disorders) | 1 | 1
Crying spells (Psychiatric disorders) | 1 | 1
Hyperactivity (Psychiatric disorders) | 2 | 1
Increased appetite (General disorders) | 1 | 1
Increased anxiety (Psychiatric disorders) | 2 | 0
Lethargy (Psychiatric disorders) | 2 | 0
Increased burping (Gastrointestinal disorders) | 3 | 0
Abnormal platelet count (Investigations) | 1 | 1
Abnormal WBC count (Investigations) | 1 | 2
SGPT outside of reference range (Investigations) | 1 | 4
SGOT outside of reference range (Investigations) | 1 | 0
TSH outside of reference range (Investigations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No